CLINICAL TRIAL: NCT00381433
Title: Pharmacokinetic Study of AVI-4065 in Cerebral Spinal Fluid Among Healthy Adult Males Following Subcutaneous Administration
Brief Title: Pharmacokinetic Study of a Single Dose of AVI-4065 in Cerebral Spinal Fluid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVI-4065-21c
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Encephalitis
Keywords: HCV; Hepatitis C virus
MeSH Terms: conditions — Encephalitis; Hepatitis C

INTERVENTIONS:
Drug: AVI-4065 Injection

SUMMARY:
AVI-4020 Injection, a phosphorodiamidate Morpholino oligomer (PMO), was found to cross the blood-brain barrier during a study of patients with presumptive West Nile virus disease. AVI-4065, which was designed to target HCV, is also a PMO; its ability to cross the blood-brain barrier is unknown. In this study, a single dose of AVI-4065 will be subcutaneously injected, and samples collected to determine if this drug crosses the blood-brain barrier. If it does, then additional investigations could be performed in people with severe forms of HCV disease in which the brain is affected.

DETAILED DESCRIPTION:
AVI-4020 Injection, a phosphorodiamidate Morpholino oligomer (PMO), was found to cross the blood-brain barrier during a study of patients with presumptive West Nile virus disease. AVI-4065, which was designed to target HCV, is also a PMO; its ability to cross the blood-brain barrier is unknown. As the incidence of HCV disease has grown, the knowledge base of this disease has likewise increased.

Encephalopathy is a recognized consequence in some patients with HCV infection. In this study, a single dose of AVI-4065 will be subcutaneously injected, and samples collected to determine if this drug crosses the blood-brain barrier. If it does, then additional investigations could be performed in people with HCV disease in which the brain is affected.

ELIGIBILITY:
Inclusion Criteria:

* Adult males 18 years to 64 years of age;
* Good general health (as evidenced by no chronic conditions, normal physical exam, vital signs within normal limits; laboratory evaluations within normal range)
* Signed and dated written informed consent form; and
* Willing to participate in all study activities and all requirements, including effective contraception (viz., a double-barrier method) during the 7-day study surveillance period.

Exclusion Criteria:

* Hematology, serum chemistry (exclusive of electrolytes), and urinalysis laboratory test values >2 times upper limits of normal or anemia (hemoglobulin <11 g/dL), leukopenia (total white blood count <3,000/µL or total neutrophils <1,500/ µL) or thrombocytopenia (platelets <100,000/µL). Electrolytes and coagulation values exceeding normal ranges are to be excluded.
* Body Mass Index (BMI) >35.
* Calculated creatinine clearance (by the Cockroft and Gault Formula) <70 mL/min, based on age and gender.
* Positive HIV-1 or HIV-2 serology.
* Positive HCV serology and/or positive plasma HCV-RNA status.
* Positive HBsAg or HBcAb status.
* Solid or hematopoetic organ transplant recipient.
* Active illness or recent illness within 30 days of the first dose of study drug.
* History of any of the following: brain injury, neoplasm, chronic or migraine headaches, cancer, meningitis or hydrocephalus.
* Usage of any prescribed, over-the-counter or illicit drug(s) within 30 days of study drug administration. Use of herbal remedies and/or supplements at the discretion of the Investigator.
* Unwilling to practice effective contraception during the study period.
* Participation in any clinical interventional trial within the previous 6 months.
* Positive drug urine screen.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2006-09; Primary Completion 2006-10 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To determine if the study drug penetrates the blood brain barrier following a single intravenous dose, and if so, the associated CSF, plasma and urine pharmacokinetics.

SECONDARY OUTCOMES:
Safety
Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Paula M Shaw, MD, Principal Investigator — NW Kinetics
Locations (1):
- NW Kinetics, Tacoma, Washington, United States